CLINICAL TRIAL: NCT04699799
Title: Characterization of Human Olfactory Amygdala Subregions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Christina Zelano, Assistant Professor, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STU00201349
Record Dates: First submitted 2021-01-04; First posted 2021-01-07 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Human Olfactory Amygdala

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- record brain activity while smelling odors (Experimental): Record brain activity while smelling odors
  Interventions: Other: Present odors to participants while recording brain activity

INTERVENTIONS:
Other: Present odors to participants while recording brain activity — Present odors to participants while recording brain activity

SUMMARY:
We aim to better understand the subregions of the human amygdala that receive direct projections from the olfactory bulb

DETAILED DESCRIPTION:
Specific Aims:

The human amygdala is part of primary olfactory cortex, in that it receives direct monosynaptic input from the olfactory bulb1-4. This suggests an important role for the amygdala in olfactory processing, yet the anatomical and functional properties of olfactory inputs to the human amygdala are largely unexplored. The overarching goal of this proposal is to elucidate the role of amygdala subregions in human olfactory processing.

The olfactory bulb projects in parallel to multiple cortical areas, each of which is thought to play a unique role in olfactory processing5-10. Within the amygdala, several distinct subregions receive direct, monosynaptic bulb input, suggesting distinct roles, yet their olfactory functions are not fully understood. Rodent studies have begun to explore potential roles for these subregions in olfactory-guided social and approach/avoid behaviors11- 15, with the first-ever recordings of the posterolateral cortical amygdala accomplished recently16. However, our understanding of these areas is still incomplete. Notably, most rodent studies on the olfactory amygdala subregions have focused on the accessory olfactory system, which humans lack. Furthermore, most human studies have not considered olfactory amygdala subregions separately17-21. This is a critical consideration, both because the majority of amygdala subregions do not receive olfactory inputs and because those that do likely play distinct roles in olfactory processing. These roles cannot be understood without analyzing the subregions separately. Thus, there is a strong need for more research into the role of the human amygdala subregions in olfaction. Importantly, olfactory amygdala subregions have been implicated in SUDEP22-26, the leading cause of death in temporal lobe epilepsy. Understanding the anatomical and functional properties of these regions is therefore of clinical importance as well.

This research will study human olfactory amygdala subregions using a multi-faceted, rigorous approach. It will combine specialized high-resolution diffusion-weighted imaging, high-resolution amygdala-targeted fMRI, rare direct electrical stimulation of the human amygdala (purely clinically prescribed) and human psychophysics, each suited to address a different question.

Aim 1: To anatomically and functionally characterize the primary olfactory cortical regions of the human amygdala. Experiments for this aim will carefully characterize human primary olfactory amygdala subregions at the anatomical and functional levels. Experiment 1A will use specialized diffusion- weighted imaging to localize olfactory tracts projecting to and from amygdala subregions. Experiment 1B will use resting fMRI and k-means clustering algorithms to parcellate and characterize amygdala subregions based on distinct whole-brain functional connectivity profiles. Experiment 1C will use event-related fMRI to functionally localize odor-responsive subregions of the amygdala. The hypothesis is that the medial, cortical and periamygdaloid subregions of the amygdala will exhibit structural connectivity with the olfactory bulb, enhanced odor-responsiveness compared to other subregions, and distinct whole-brain functional connectivity profiles.

Aim 2: To test the hypothesis that activity in distinct amygdala subregions reflects distinct olfactory behaviors. Experiments for this aim will use fMRI-derived ensemble patterns and time-series to explore distinct olfactory roles for amygdala subregions, with excellent spatial resolution and simultaneous coverage of the entire amygdala. The use of fMRI ensemble patterns is ideal, since olfactory cortical areas including the amygdala use a distributive mode of coding16. Experiment 2A will use fMRI to measure activity across all amygdala subregions while presenting identical odors under different ecologically relevant contexts (social, spatial and food). Experiment 2B will use fMRI to examine correlations between amygdala fMRI patterns and olfactory approach/avoid behaviors. The hypothesis is that, as in rodents, activity in the medial amygdala will reflect olfactory-guided social perceptual decisions and that activity in the cortical amygdala will reflect olfactory-guided approach/avoid behaviors.

Aim 3: To assess the necessity of olfactory amygdala subregions in distinct olfactory behaviors. To assess the necessity of olfactory amygdala subregions in the distinct olfactory behaviors described above in Aim 2, Experiment 3 will use intracranial electrophysiology methods to record directly from, and deliver electrical stimulation directly into, human olfactory amygdala sub-regions during the olfactory tasks from Aim 2. Stimulation will not deviate from clinical protocols, and will be performed by clinicians only. This method provides direct recordings of neural activity, and allows disruption of neural activity to test the necessity of specific regions for particular behaviors. The hypothesis is that disruption of oscillatory activity in the cortical amygdala will disrupt olfactory approach/avoid behaviors, while disruption of oscillatory activity in the medial amygdala will disrupt olfactory social perceptual decisions.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years of age

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Strength of olfactory input to amygdala subregions | 4 years
  We will assess the quantity of input to each amygdala subregion from the olfactory tract

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern human olfaction lab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
All data will be made freely available on our lab website and/or GitHub page. All raw data will be available
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Some of the above may be made available on our lab website, if relevant for the particular study. Data will be available with no time limitations. Data will be made available once published.

DOCUMENTS (1):
  • Informed Consent Form (2023-03-20): https://cdn.clinicaltrials.gov/large-docs/99/NCT04699799/ICF_001.pdf